CLINICAL TRIAL: NCT04879004
Title: Effectiveness of Bilateral Erector Spinae Plane Block (ESPB) in Laparoscopic Colectomies -A Randomized, Controlled, Double Blind, Prospective Trial
Brief Title: EFFECT - EFFectiveness of ESPB (Erector Spinae Plane Block) in Laparoscopic Cοlectomies Trial
Acronym: EFFECT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Democritus University of Thrace (Other)
Collaborators: Aristotle University Of Thessaloniki (Other)
Responsible Party: Principal Investigator, Freideriki Sifaki, M.D., Msc, Democritus University of Thrace
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 1147/7.10.2019
Record Dates: First submitted 2021-05-01; First posted 2021-05-10 (Actual); Last update posted 2021-05-10 (Actual); Status verified 2021-05

CONDITIONS: Pain, Postoperative; Acute Pain; Postoperative Complications; Pain; Ropivacaine; Analgesia; Regional Anesthesia; Analgesics; Anesthesia, Local; Colorectal Cancer; Perioperative Pain
Keywords: Erector Spinae Plane Block; Regional Anaesthesia; Opioid - Free Anaesthesia; Opioid Sparing Techniques; Laparoscopic Colectomy; Perioperative Pain; General Surgery
MeSH Terms: conditions — Pain, Postoperative; Acute Pain; Postoperative Complications; Pain; Agnosia; Colorectal Neoplasms | interventions — Ropivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Ropivacaine Group (Experimental): ESPB performed with infusion of Ropivacaine 0,375% (20 ml at ech side)
  Interventions: Drug: Ropivacaine injection
- Control Group (Placebo Comparator): ESPB performed with infusion of N/S 0,9% (20 ml at each side)
  Interventions: Drug: Ropivacaine injection

INTERVENTIONS:
Drug: Ropivacaine injection — Effect of continuous ESPB performed with Ropivacaine 0,375% infusion, in patients undergoing elective laparoscopic colectomy.

SUMMARY:
The aim of the trial is to study the efficacy of continuous bilateral Erector Spinae Plane Block (ESPB) in managing perioperative pain in patients who undergo elective laparoscopic colectomy.

DETAILED DESCRIPTION:
Laparoscopic colectomy is a common surgery performed by general surgeons for a variety of reasons, such as colon cancer, inflammatory bowel disease, multiple precancerous colon polyps. Nowadays, due to the evolution of laraposcopic techniques, laparoscopic colectomies are performed with minimally invasive procedures. However, most patients complain for moderate to severe post-operative pain, which requires the application of multimodal analgesia recipes and the administration of large doses of opioids perioperatively, in order to be relieved. Due to the opioid crisis observed in the U.S. and in many european countries and due to the variety of adverse effects observed after the administration of opioids (respiratory depression, nausea, vomiting, delayed mobilization of gastrointestinal system and the patient), which augment not only the hospitalization time but also the hospitilization cost of the patients, anesthesiologists tend to limit their administration, especially in colectomies.

Erector Spinae Plane Block (ESPB) is an innovating trunk block, which was first described in 2016 by Forrero et. al in order to relieve neuropathic pain. Since then, it was embraced by modern anesthesia practices and is currently effectively performed for chronic pain, acute post-traumatic and acute post-operative pain, in various surgical procedures. Specifically, ESPB has been performed for the treatment of thoracic neuropathic pain, of acute post-operative pain after thoracotomy, laparoscopic cholecystectomy, total hip arthroplasty, modified radical mastectomy, emergent laparotomy and after various surgical procedures of the spine, with good results.

There are no clinical trials that study the effectiveness of continuous bilateral Erector Spinae Plane Block in laparoscopic colectomies.

This trial is a randomized, controlled, double - blind, prospective trial, predominantly aiming at evaluating the effectiveness of continuous bilateral Erector Spinae Plane Block (ESPB) in managing perioperative pain in patients who undergo elective laparoscopic colectomy.

This trial will recruit 40 patients (men and women), aged 18 to 85 years old who will undergo laparoscopic colectomy, performed by the same experienced, surgical team.

Patients will be randomized into two groups, Group B (Block Group - Ropivacaine 0,375%) and Group C (Control group - N/S 0,9%).

ESPB will be performed bilaterally, accompanied with the placement of catheters for continuous solution infusion, by the same, experienced in regional anesthesia anesthesiologist, before the induction of general anesthesia. The solutions administered during the performance of ESPB, will be prepared by an independent anesthesiology nurse. The quality of the ultrasound image and the pain intensity during the performance of ESPB, as well as the dermotomes blocked by ESPB and the complications that may arise after the performance of the block, will be recorded.

The age, sex, Body Mass Index and American Society of Anesthesiologists (ASA) classification of the participants, will be recorded. Preoperative standard laboratory tests, as well as TNF-a, Interleukine-1 and Interleukine-6 levels will be recorded.

After the induction of general anesthesia [propofol (2,5 mg/kg), fentanyl (1 γ/kg), rocuronium (0,6 mg/kg)], general anesthesia will be maintained with desflurane titration, guided by BIS Monitor readings. In all patients, remifentanil infusion will be titrated in order to achieve intraoperative analgesia, guided by Nociception Monitoring (NOL Monitor). In all patients Magnesium Sulphate 50 mg/kg and Pantoprazole 40 mg will be administered at the start of the surgical procedure. Paracetamol 1000 mg, Tramadol 100 mg, Droperidol 1,25 mg and Ondansetron 4 mg will be also administered to all patients 30 minutes before the end of surgery. During surgery, vital signs, BIS and NOL readings, Cardiac Output, Stroke Volume Variation, Glucose and Lactate levels will be recorded. Total fluids, desflurane and remifentanyl administration, urine output, as well as the administration of other drugs will also be recorded. At the end of surgery, Train of Four stimulation will be performed and in the presence of remaining neuromuscular blockade, sugammadex will be administered in the proper doses.

In all patients, post - operative analgesia will include administration of Paracetamol 1000 mg every 6 hours. Tramadol 50 mg will be offered as rescue analgesia, if NRS pain score of the patient is > 4. 12, 24, 36 and 48 hours after the performance of ESPB, Ropivacaine 0,375% (patients randomized in Group B) or N/S 0,9% (patients randomized in Group C) will be infused through the ESPB catheters.

The duration of stay of the patient in Post Anesthesia Care Unit (PACU), the Aldrete Score and the vital signs the moment the patient leaves the PACU, will be recorded.

Post - operative observation of the patient will include recording of NRS pain score at rest and activity, Post-Operative Nausea and Vomiting Score, tramadol consumption, vital signs, 12, 24, 36, 48, 60, 72, 84 and 96 hours after the end of surgery. Quality of Recovery Score of the patient will be recorded 72 hours after the end of surgery. Mobilization time of the patient and of the gastrointestinal tract, the time of removal of bladder catheter and drainages, the time of start of oral fluids and enteral nutrition, the discharge time and the total cost, will also be recorded. The satisfaction score of the patient in a scale from 1 to 6, 96 hours after the end of surgery will be recorded. Standard laboratory tests of the first, second and third post-operative days will be recorded, as well as the TNF-a, Interleukine-1 and Interleukine-6 levels the first and the fourth post-operative day.

ELIGIBILITY:
Inclusion Criteria:

ASA I, II, III Laparoscopic colectomy Elective surgery

Exclusion Criteria:

Patient refusal Known allergies to local anesthetics Other contraindications to regional anesthesia Infection or anatomic anomalies on injection site Uncontrolled hypertension Severe liver or kidney disease Pregnancy Known depression or psychiatric disorders, dementia Drug or alcohol abuse Inadequate command of Greek language

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-05-31 (Estimated); Study Completion 2022-05-31 (Estimated)

PRIMARY OUTCOMES:
Total Perioperative Tramadol Consumption | 96 hours after surgery
  Total Perioperative Tramadol Consumption
Quality of Recovery | 72 hours Post - Operatively
  Quality of Recovery-15 [(QoR) -15] Questionnaire. A questionnaire which consists of 15 questions in two Parts, rated from 0 to 10 ("0" is the worst and "10" is the best answer). The worst overall score is 0 and the best overall score is 150.
Mobilization Time | In a time frame of up to 72 hours Post - Operatively
  Time of Mobilization of the gastrointestinal tract and of the patient
Start of Oral Fluids and Nutrition | In a time frame up to 72 hours Post - Operatively
  Time of start of oral fluids and enteral nutrition
Satisfaction from Perioperative Analgesia | 96 hours post - operatively
  Satisfaction Score of the patient regarding perioperative analgesia, using a numerical rating scale from 1 to 6, where "1" means not satisfied at all and "6" means completely satisfied.
Hospitalization Days | In a time frame up to 2 Weeks Post - Operatively
  Duration of hospital stay after surgery in days

SECONDARY OUTCOMES:
Pain Score, Post Operative Nausea and Vomiting Score at discharge from Post-Anesthesia Care Unit (PACU) | Immediately Post - Operatively
  Pain score at discharge from Post-Anesthesia Care Unit (PACU), ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable", Post Operative Nausea and Vomiting Score at discharge from Post-Anesthesia Care Unit (PACU), ranging from 0 to 2, where "0" means no PONV, "1" means nausea and "2" means vomiting.
Pain Score, Post Operative Nausea and Vomiting Score 12 hours post-operatively | 12 hours post - operatively
  Pain score 12 hours post - operatively, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable", Post Operative Nausea and Vomiting Score 12 hours post - operatively, ranging from 0 to 2, where "0" means no PONV, "1" means nausea and "2" means vomiting.
Pain Score, Post Operative Nausea and Vomiting Score 24 hours post-operatively | 24 hours post - operatively
  Pain score 24 hours post - operatively, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable", Post Operative Nausea and Vomiting Score 24 hours post - operatively, ranging from 0 to 2, where "0" means no PONV, "1" means nausea and "2" means vomiting.
Pain Score, Post Operative Nausea and Vomiting Score 36 hours post-operatively | 36 hours post - operatively
  Pain score 36 hours post - operatively, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable", Post Operative Nausea and Vomiting Score 36 hours post - operatively, ranging from 0 to 2, where "0" means no PONV, "1" means nausea and "2" means vomiting.
Pain Score, Post Operative Nausea and Vomiting Score 48 hours post-operatively | 48 hours post - operatively
  Pain score 48 hours post - operatively, ranging from 0 to 10, where 0 means "no pain" and 10 means "worst pain imaginable", Post Operative Nausea and Vomiting Score 48 hours post - operatively, ranging from 0 to 2, where "0" means no PONV, "1" means nausea and "2" means vomiting.
Total Desflurane Consumption | Intra - Operatively
  Total intraoperative Desflurane Consumption
Total Remifentanyl Consumption | Intra - Operatively
  Total intraoperative Remifentanyl Consumption
Post Anesthesia Care Unit (PACU) Duration of stay | Immediately post-operatively
  Duration of patient stay at PACU
Total Cost | Perioperatively
  Total cost of surgery, anesthesia and hospitalization
TNF-a, IL-1, IL-6 levels post-operatively | Pre-operatively and the 1st and 4th day post-operatively
  Comparison of TNF-a, Interleukine-1 and Interleukine-6 levels preoperatively and post - operatively (the first and fourth day after surgery)

CONTACTS AND LOCATIONS:
Locations (1):
- Georgios Papanikolaou, General Hospital of Thessaloniki, Thessaloniki, Thessaloniki, Greece

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Kwon HM, Kim DH, Jeong SM, Choi KT, Park S, Kwon HJ, Lee JH. Does Erector Spinae Plane Block Have a Visceral Analgesic Effect?: A Randomized Controlled Trial. Sci Rep. 2020 May 21;10(1):8389. doi: 10.1038/s41598-020-65172-0. PMID 32439926
- [Background] Tulgar S, Selvi O, Senturk O, Serifsoy TE, Thomas DT. Ultrasound-guided Erector Spinae Plane Block: Indications, Complications, and Effects on Acute and Chronic Pain Based on a Single-center Experience. Cureus. 2019 Jan 2;11(1):e3815. doi: 10.7759/cureus.3815. PMID 30868029
- [Background] Beck DE, Margolin DA, Babin SF, Russo CT. Benefits of a Multimodal Regimen for Postsurgical Pain Management in Colorectal Surgery. Ochsner J. 2015 Winter;15(4):408-12. PMID 26730224
- [Background] Gustafsson UO, Scott MJ, Schwenk W, Demartines N, Roulin D, Francis N, McNaught CE, Macfie J, Liberman AS, Soop M, Hill A, Kennedy RH, Lobo DN, Fearon K, Ljungqvist O; Enhanced Recovery After Surgery (ERAS) Society, for Perioperative Care; European Society for Clinical Nutrition and Metabolism (ESPEN); International Association for Surgical Metabolism and Nutrition (IASMEN). Guidelines for perioperative care in elective colonic surgery: Enhanced Recovery After Surgery (ERAS((R))) Society recommendations. World J Surg. 2013 Feb;37(2):259-84. doi: 10.1007/s00268-012-1772-0. No abstract available. PMID 23052794
- [Background] Benyamin R, Trescot AM, Datta S, Buenaventura R, Adlaka R, Sehgal N, Glaser SE, Vallejo R. Opioid complications and side effects. Pain Physician. 2008 Mar;11(2 Suppl):S105-20. PMID 18443635
- [Background] Forero M, Adhikary SD, Lopez H, Tsui C, Chin KJ. The Erector Spinae Plane Block: A Novel Analgesic Technique in Thoracic Neuropathic Pain. Reg Anesth Pain Med. 2016 Sep-Oct;41(5):621-7. doi: 10.1097/AAP.0000000000000451. PMID 27501016
- [Background] De Cassai A, Cin SD, Zarantonello F, Ban I. Erector spinae plane block as a rescue therapy for uncontrolled pain after laparotomic surgery: A report of two cases. Saudi J Anaesth. 2019 Jan-Mar;13(1):66-68. doi: 10.4103/sja.SJA_449_18. PMID 30692892